CLINICAL TRIAL: NCT00217984
Title: Intensive Intervention for Smokers in Alcohol Treatment
Brief Title: Intensive Intervention for Smokers - 6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-09253-6; P50DA009253 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Tobacco Use Disorder; Alcohol Dependence
Keywords: Tobacco use disorder; Alcohol dependence
MeSH Terms: conditions — Tobacco Use Disorder; Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive intervention (Experimental): Extended cognitive behavior therapy (16 sessions) plus nicotine patches and lozenges
  Interventions: Behavioral: Extended cognitive behavior therapy
- Usual care (Other): Referral to the smoking cessation clinic
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — Referral to smoking cessation clinic
  Other Names: Smoking cessation clinic
  Arms: Usual care
Behavioral: Extended cognitive behavior therapy — 16 sessions of cognitive behavior therapy over 6 months
  Arms: Intensive intervention

SUMMARY:
The purpose of this study was to determine the efficacy and cost-effectiveness of an intensive smoking cessation intervention that utilizes extended cognitive-behavioral therapy and combination nicotine replacement (CNR) in a randomized controlled trial. The intensive intervention was compared to usual care involving referral to a free-standing smoking cessation program that provides brief counseling and CNR. We recruited 162 smokers, ages 18 to 75, who are enrolled in the Drug and Alcohol Treatment (DAT) programs at the San Francisco VA Medical Center (SFVAMC) and Santa Rosa VA Community-based Outpatient Clinic (CBOC). To be eligible, participants had to be abstinent from alcohol for at least one week, but not more than 30 days. We compared outcomes for the two study arms by assessing biochemically-validated point-prevalence smoking status at 3, 6, 9, and 12 months post-baseline and continuous abstinence over the 12-month follow-up. Expired-air carbon monoxide (CO) was used to biochemically verify 7-day point prevalence abstinence. We also conducted an economic analysis to determine the cost-effectiveness of the intensive intervention compared with usual care. We also examined cross-relapse patterns during the follow-up period, assessing changes in mood states and use of tobacco, alcohol, and other drugs at 3, 6, 9, and 12 months.

DETAILED DESCRIPTION:
Introduction. The purpose of this study was to investigate the efficacy of an intensive tobacco cessation intervention for alcohol-dependent smokers in early recovery.

Methods. A total of 162 alcohol-dependent smokers were randomized to either intensive intervention for smoking cessation or usual care. The intensive intervention consisted of 16 sessions of individual cognitive behavior therapy (CBT) and combination nicotine replacement therapy that lasted 26 weeks. Usual care involved referral to a free-standing smoking cessation program that provided smoking cessation counseling of varying duration and guideline-concordant medications. The primary cessation outcome was verified 7-day point prevalence abstinence (PPA) at 12, 26, 38, and 52 weeks.

Results. At 12 and 26 weeks, the verified 7-day point-prevalence quit rate was significantly higher for the intensive intervention group than for the usual care group (both p = .03). However, the quit rates for the two treatment groups were not significantly different at 38 or 52 weeks. Verified 30-day alcohol abstinence rates were not significantly different for the two treatment groups at any of the follow-up assessments.

Conclusions. The intensive smoking cessation intervention yielded a higher short-term smoking quit rate without jeopardizing sobriety. A chronic care model might facilitate maintenance of smoking cessation during the first year of alcohol treatment and perhaps for longer periods of time. It is hoped that studies such as this will inform the development of more effective interventions for concurrent alcohol and tobacco use disorders.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* alcohol as primary drug of abuse
* currently smoking at least 10 or more cigarettes
* abstinent from alcohol for at least 7 days and not more than 30 days
* self-reported interest in quitting smoking

Exclusion Criteria:

* any contraindications for nicotine patches or lozenges (e.g., unstable angina or recent myocardial infarction
* skin allergy to the nicotine patch
* severe cardiovascular disease
* lactation
* pregnancy by self-report or by positive serum pregnancy test in pre-menopausal women)
* unstable psychiatric disorder
* severe cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-07; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
7 day point prevalence of cigarette abstinence | Assessed at 3, 6, 9, and 12 months
  Participants are asked whether they smoked any cigarettes during the past seven days. Expired-air carbon monoxide is measured to validate abstinence.

SECONDARY OUTCOMES:
Alcohol use | Assessed at 3, 6, 9, and 12 months
  Participants were asked to report use of alcohol during the past 90 days, using a timeline follow-back interview method

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Carmody, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- VA Medical Center, San Francisco, California, United States